CLINICAL TRIAL: NCT07142278
Title: A Phase 1 Study of the Safety and Tolerability of DUVAX, a Dual-Target Alzheimer's Vaccine (Amyloid-Beta and Tau), in Healthy Volunteers
Brief Title: DUVAX: A Phase 1 Alzheimer's Vaccine Study Targeting Amyloid-Beta and Tau
Acronym: DU-PRISM
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nuravax, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Institute for Molecular Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DUVAX-101; 1R44AG091903 (NIH)
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease; Alzheimer Disease (AD); Preclinical Alzheimer's Disease
Keywords: Asymptomatic Alzheimer Disease; Preclinical Alzheimer's disease; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Parallel assignment of participants to DUVAX or placebo within two dose cohorts (200 µg and 400 µg). Each cohort will be randomized 3:1 (DUVAX: placebo), with sentinel participants enrolled first for safety review before the full cohort is enrolled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, study staff, care providers, and outcomes assessors will remain blinded to treatment allocation. The investigational product and placebo are identical in appearance, packaging, and administration. Randomization codes will be maintained by an unblinded pharmacist or designee and will not be disclosed until study unblinding, except in case of medical emergency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active - DUVAX 200 µg (Experimental): Participants receive three intramuscular injections of DUVAX 200 µg formulated with Adjuvant at Weeks 0, 4, and 22.
  Interventions: Biological: DUVAX 200 µg
- Active - DUVAX 400 µg (Experimental): Participants receive three intramuscular injections of DUVAX 400 µg formulated with Adjuvant at Weeks 0, 4, and 22.
  Interventions: Biological: DUVAX 400 µg
- Placebo (Adjuvant only) (Placebo Comparator): Participants receive three intramuscular injections of placebo (adjuvant formulation without active antigen) at Weeks 0, 4, and 22.
  Interventions: Biological: Placebo (Adjuvant only)

INTERVENTIONS:
Biological: DUVAX 200 µg — Intramuscular injection of 200 µg DUVAX formulated with Adjuvant, administered at Weeks 0, 4, and 22
  Arms: Active - DUVAX 200 µg
Biological: DUVAX 400 µg — Intramuscular injection of 400 µg DUVAX formulated with Adjuvant, administered at Weeks 0, 4, and 22
  Arms: Active - DUVAX 400 µg
Biological: Placebo (Adjuvant only) — Intramuscular injection of placebo consisting of Adjuvant formulation in phosphate-buffered saline without active antigen, administered at Weeks 0, 4, and 22
  Arms: Placebo (Adjuvant only)

SUMMARY:
This Phase 1 study will test the safety and immune response of the investigational vaccine DUVAX in healthy adults. Participants will be randomly assigned to receive either DUVAX or placebo by intramuscular injection. The study will evaluate how well the vaccine is tolerated and whether it produces antibodies against Alzheimer's disease-related proteins.

DETAILED DESCRIPTION:
This is a first-in-human, randomized, double-blind, placebo-controlled Phase 1 trial of DUVAX, an adjuvanted vaccine, in up to 24 healthy participants aged 40-65 years. Two dose levels (200 µg and 400 µg) will be evaluated. Participants will receive three intramuscular doses at Weeks 0, 4, and 22, with safety and immunogenicity monitoring through one year after the last vaccination.

The primary objective is to assess safety and tolerability. The secondary objective is to measure immunogenicity by evaluating antibody responses against amyloid beta (Aβ) and tau proteins.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and non-pregnant, non-lactating females, 40-65 years old
* BMI between 18.0 and 32.0 kg/m²
* Medically healthy with no significant abnormalities in medical history, exam, labs, ECG, or MRI
* Signed informed consent
* Women of childbearing potential: negative pregnancy test and use of effective contraception
* Men: vasectomized or agree to use condoms / not donate sperm during the study period

Exclusion Criteria:

* Clinically significant medical or psychiatric illness that may affect safety or study results
* MRI abnormalities (e.g., infarcts, microbleeds, ARIA-E) or contraindications to MRI
* Significant lab abnormalities (e.g., liver, kidney, hematology) or positive HIV/HBV/HCV tests
* Uncontrolled blood pressure, abnormal heart rate, or prolonged QTc interval
* Recent serious illness, surgery, or investigational drug use within 30 days
* Prior amyloid-beta or tau immunotherapy within 1 year
* Use of immunosuppressive agents or chronic anticoagulants
* History of severe vaccine reactions, autoimmune disease, or significant allergies

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Participants with Treatment-Emergent Adverse Events (TEAEs), including Adverse Events of Special Interest (AESI) | From baseline (Day 1) through Week 74 (end of study follow-up)
  Safety will be assessed by recording the number and type of treatment-emergent adverse events (TEAEs), including adverse events of special interest (AESI), reported from baseline through the follow-up period. Events will be summarized by severity and relationship to study treatment.

SECONDARY OUTCOMES:
Serum anti-Aβ antibody titers (IgM, IgG, and IgG subclasses) | Baseline, Weeks 2, 4, 6, 22, 25, and 38
  Immunogenicity will be assessed by measuring antibody titers against amyloid-beta (Aβ), including total IgM, total IgG, and IgG subclasses (IgG1, IgG2, IgG3, IgG4). Changes from baseline will be compared.

OTHER OUTCOMES:
Serum anti-Tau antibody titers (IgM, IgG, and IgG subclasses) | Baseline, Weeks 2, 4, 6, 22, 25, and 38
  Immunogenicity will be assessed by measuring antibody titers against tau protein, including total IgM, total IgG, and IgG subclasses (IgG1, IgG2, IgG3, IgG4). Changes from baseline will be compared.
Serum anti-MultiTEP antibody titers (IgM, IgG, and IgG subclasses) | Baseline, Weeks 2, 4, 6, 22, 25, and 38
  Immunogenicity will be assessed by measuring antibody titers against MultiTEP carrier epitopes, including total IgM, total IgG, and IgG subclasses (IgG1, IgG2, IgG3, IgG4). Changes from baseline will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Anahit Ghochikyan, PhD, Principal Investigator — IMM; David Cribbs, PhD, Principal Investigator — Nuravax, Inc.; Roman Kniazev, Study Chair — Nuravax, Inc.
Locations (1):
- Palm Springs Community Health Center, Miami Lakes, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying published results (demographics, outcomes, and adverse events) will be shared.
Time Frame: At the time of primary publication or within 9 months of database lock, whichever occurs first.
Access Criteria: Available to qualified researchers upon request and subject to review by the study investigators.